CLINICAL TRIAL: NCT05014646
Title: Phase 2 Trial of Leflunomide in African-American and European-American Patients With High-Risk Smoldering Multiple Myeloma
Brief Title: Leflunomide for the Treatment of High-Risk Smoldering Multiple Myeloma in African-American and European-American Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21049; NCI-2021-07263 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21049 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Cholestyramine Resin; Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (leflunomide) (Experimental): Patients receive leflunomide PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cholestyramine; Drug: Leflunomide

INTERVENTIONS:
Drug: Cholestyramine — Given PO
  Other Names: Cholybar; Colestyramine; Duolite AP143 Resin; Questran; Questran Light
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101

SUMMARY:
This phase II trial studies the effects of leflunomide in treating African-American and European-American patients with high-risk smoldering multiple myeloma. Leflunomide is used to decrease the body's immune response and may delay the symptoms of multiple myeloma in patients of African-American and European decent.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-myeloma activity of leflunomide, when given as a single agent, as assessed by freedom from progression at 2-years.

II. To evaluate the safety and tolerability of single agent leflunomide.

SECONDARY OBJECTIVES:

I. To summarize and assess toxicities by type, frequency, severity, attribution, time course and duration.

II. To estimate overall and progression-free survival probabilities. III. To estimate response rate and duration of response. IV. To describe the impact of treatment on quality of life, as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score version (v)3.0.

EXPLORATORY OBJECTIVES:

I. To characterize the molecular evolution of the tumor cells. II. To evaluate whether specific genetic subtypes respond differently to leflunomide.

III. To evaluate the role of immune cells in the progression of smoldering multiple myeloma (SMM).

IV. To evaluate the role of leflunomide in modulating the immune system. V. To examine the relationship between immunological changes and disease progression.

OUTLINE:

Patients receive leflunomide orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up yearly.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients must be age >= 18 years
* Patients must have a life expectancy of > 24 months
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must identify as African-American OR European-American
* Patients must have a diagnosis of high risk smoldering multiple myeloma, as defined below:

  * The presence of >= 2 of the following risk factors:

    * Bone marrow plasma cell percentage (BMPC%) > 20%
    * Serum M-protein > 2 g/dL
    * Free light chain ratio (FLCr) > 20
* A diagnosis of high-risk SMM must have been made within the last 3 years
* At least 2 weeks from prior therapy to time of start of treatment. Prior therapy includes steroids (except prednisone or equivalent - up to 10 mg per day is allowed)
* Platelet count >= 50,000/uL. Platelet transfusions are not allowed within 14 days of platelet assessment
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.0 x upper limit of normal (ULN)
* Total bilirubin < 1.5 x ULN
* Calculated creatinine clearance (CrCl) >= 30 mL/min per 24-hour urine collection or the Cockcroft-Gault formula
* Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only), to be performed locally within the screening period
* Negative for tuberculosis antigen (e.g. T-Spot test)
* Negative for hepatitis A, B, or C infection
* Adequate pulmonary function as defined by forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% of predicted by pulmonary function testing
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for three months following duration of study participation. The effects of study treatment on a developing fetus have the potential for teratogenic or abortifacient effects. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

  * A female of childbearing potential is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months

Exclusion Criteria:

* Prior treatment with leflunomide
* Prior treatment for smoldering multiple myeloma
* Current or planned use of other investigational agents, or concurrent biological, chemotherapy, or radiation therapy during the study treatment period. Current or planned growth factor or transfusion support until after initiation of treatment. If growth factor or transfusion support is provided between screening and start of treatment, the participant will no longer be eligible
* Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

  * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  * Renal insufficiency: creatinine clearance < 30 mL per min or serum creatinine > 177 umol/L (> 2 mg/dL)
  * Anemia: hemoglobin value of > 20 g/L below the lower limit of normal, or a hemoglobin value < 10 g/dL
  * Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography (PET)-CT
* Any one or more of the following biomarkers of malignancy:

  * Clonal bone marrow plasma cell percentage >= 60%
  * Involved:uninvolved serum free light chain ratio >= 100 (Involved free light chain must be >= 100 mg/L)
  * >= 1 focal lesions on magnetic resonance imaging (MRI) studies (>= 5 mm in size each)
  * Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible
* Prior diagnosis of rheumatoid arthritis
* Prior allogeneic transplant
* Acute active infection requiring systemic therapy within 2 weeks prior to enrollment
* Pre-existing liver disease
* Known human immunodeficiency virus (HIV) infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leflunomide and cholestyramine
* Non-hematologic malignancy within the past 3 years aside from the following exceptions:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Prostate cancer < Gleason grade 6 with a stable prostate specific antigen (PSA)
  * Successfully treated in situ carcinoma of the breast
* Clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or the patient's ability to give informed consent
* Pregnant women and women who are lactating. Leflunomide has potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression to multiple myeloma | At 2 years
Incidence of adverse events | Up to 30 days after last dose
  Measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5. Will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, serum concentration of the active leflunomide metabolite, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Overall survival | From start of treatment to death, or last follow-up, whichever comes first, assessed up to 2 years
Progression-free survival | From randomization to progression or death or loss to follow up, whichever comes first, assessed up to 2 years
Freedom-from progression | From start of treatment to the first assessment showing symptomatic disease, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Rosenzweig, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health University City/LCI-University, Charlotte, North Carolina